CLINICAL TRIAL: NCT01957189
Title: An Open Label, Single Sequence, Three Period, Drug-Drug Interaction Study To Examine The Pharmacokinetics Of Dutasteride And Tamsulosin And Their Interactions In Chinese Male Healthy Volunteers
Brief Title: This Will be an Open-label, Three-period, Fixed-sequence Study to Evaluate the Drug-drug Interaction, Pharmacokinetics and Safety of Dutasteride and Tamsulosin When Administered Alone and In-combination in Chinese Healthy Male Volunteers. The Study Will Last Approximately Eleven Weeks. Blood Samples
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200254
Record Dates: First submitted 2013-10-04; First posted 2013-10-08 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Prostatic Hyperplasia
Keywords: pharmacokinetics, Chinese; Avodart, Duodart, dutasteride, tamsulosin, drug-drug interaction,
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dutasteride with/ without Tamsulosin (Experimental): All subjects will be assigned to the same treatment group
  Interventions: Drug: Dutasteride and Tamsulosin

INTERVENTIONS:
Drug: Dutasteride and Tamsulosin — 0.5mg dutasteride once a day on Day 1 Period A , and Day 5 Period C,0.2mg Tamsulosin once a day on Day 1 to Day 7 in Period B and Period C

SUMMARY:
This will be an open-label, three-period, fixed-sequence study to evaluate the drug-drug interaction, pharmacokinetics and safety of dutasteride and tamsulosin when administered alone and in-combination in Chinese healthy male volunteers.

DETAILED DESCRIPTION:
This will be an open-label, three-period, fixed-sequence study to evaluate the drug-drug interaction, pharmacokinetics and safety of dutasteride and tamsulosin when administered alone and in-combination in Chinese healthy male volunteers. The study will last approximately eleven weeks. Blood samples for pharmacokinetic analysis will be taken at pre-specified times. Safety will be assessed by measurement of concurrent medication,changes in clinical laboratory values, ECG, vital signs, and collection of adverse events.Approximately 24 healthy adult males will be enrolled such that approximately 18 subjects complete dosing and critical assessments.This will be an open label, single sequence, three-period study. Approximately 24 healthy male volunteers will be enrolled. At the first study period, the subjects will receive 0.5mg of dutasteride (Dut) as a single dose (SD) under fed conditions. Serum sampling will take place pre-dose and over the next 72 hours post dose (Per. A). After a 28-30 days washout, the subjects will be brought in and be given 0.2mg tamsulosin as Harnal D tablet for 7 days with the morning meal. Serum sampling for pharmacokinetics of tamsulosin will take place at day 1, day 2 and day 3 pre-dose and at days 4 for 24 hours (Per. B). On the next day (Day 5), the subjects will be given both 0.2mg tamsulosin Harnal D tablet and 0.5mg of dutasteride. Serum sampling will take place at Day 5 pre-dose and followed for 72 hours (Per. C) for both dutasteride and tamsulosin. Subjects will participate in a follow-up visit approximately 2 weeks after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Ethnic Chinese male subject between the ages of 18 and 45 years old inclusive, at the time of signing the informed consent.
* Ethnic Chinese are defined as being born in China, having four ethnic Chinese grandparents, stay in China for most time and be abroad no more than 10 years.
* Healthy subjects defined as individuals who are free from significant cardiac,pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrinological and psychiatric disease as determined by medical history,physical examination, vital signs, electrocardiogram (ECG) and clinical laboratory test results.
* Body weight >= 50 Kilogram (kg) and BMI within the range 19 - 24 kg/m2(inclusive).
* Serum creatinine < 1.5xULN at screening.
* Based on single or averaged QTc values of triplicate ECGs obtained over a brief recording period:

[QTc] < 450 Milliseconds (msec); or QTc < 480 msec in subjects with Bundle Branch Block.

* Alanine aminotransferase (ALT), alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Subjects must be able and willing to stop using of any tobacco or nicotine containing products 24 hours prior to each dose and for the duration of confinement. At the discretion of the Investigator, light smokers (smoking ≤10 cigarettes a day) would be considered for the study inclusion.
* Willing and able of giving written informed consent, which includes compliance with the all the requirements and restrictions listed in the consent form for the full duration of the study, and able to understand and follow instructions related to study procedures.
* Able to swallow and retain oral medication.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods.This criterion must be followed from the time of the first dose of study medication until 50 days after the last dose.

Exclusion Criteria:

* The subject has received an investigational product or participated in any other research trial within 6 months or 5 half-lives, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of current study medication or anytime during the study period, or exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Previous use of the following medications or involvement in an investigational drug study of any of these in the previous three months prior to screening:

finasteride, (PROSCAR, PROPECIA) investigational 5 ARIs (i.e., GI198745 and epristeride) phytotherapy (i.e., over the counter plant extracts for BPH and alopecia) anabolic steroids (i.e., oxandrolone, testosterone ester) drugs with anti-androgenic properties (i.e., spironolactone, cimetidine) alpha-1 antagonists (i.e., terazosin, doxazosin, alfuzosin and tamsulosin) antihypertensive agents or diuretics

* Previous donation of blood or blood products in excess of 500 mL within a 90 day prior to the first dose of investigational products and the subject agrees not to donate blood during this study.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >21 units for males. One unit is equivalent to 8 g of alcohol: a half-pint (~240 ml) of beer, 1 glass (125 ml) of wine or 1 (25 ml) measure of spirits. Subjects must be able and willing to abstain from beverages and foods containing alcohol 24 hours prior to the first dose of study medication and until collection of the final pharmacokinetic sample during each period.
* Positive test result for Hepatitis B surface antigen (HBsAg), Hepatitis C surface antibody (HCAb), or HIV antibody at Screening.
* Subjects with a positive urinary drug or alcohol screen at screening and at Day -1of study participation.
* Poor metabolizer for CYP2D6 substrates as determined by genotyping of selected CYP2D6 variants at screening.
* Subjects with an acute illness requiring treatment by a physician within 30 days proceeding the screening period of the study, or a significant febrile illness within five days of the first day the subject will receive the study drug.
* Subjects with sensitivity to currently available 5 ARIs (i.e., finasteride).
* Subjects with sensitivity to currently available alpha 1 antagonists (i.e., terazosin doxazosin, alfuzosin and tamsulosin). History or presence of allergy, intolerance, or contraindication to tamsulosin or dutasteride or any of its components, soya or peanuts, or drugs of these therapeutic classes, or a history of drug or other allergy (including true sulfonamide allergy) that, in the opinion of the physician responsible, contraindicates their participation.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal, dietary supplements within 7 days (or 14 days if the drug is a potential enzyme inducer, such as St. John's Wort, Black Cohosh, Dong Quai, milk thistle, and licorice) or 5 half-lives (whichever is longer) prior to the first dose of study medication and up to 4 days from receiving the last dose of study medication.
* Unable to refrain from the consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pomelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication until collection of the last blood sample for determination of pharmacokinetic parameters.
* Any clinically significant abnormality on the screening ECG or screening laboratory tests.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* History of postural hypotension, dizziness, poor hydration, vertigo, vaso-vagal reactions or any other signs and symptoms of orthostasis, which in the opinion of the investigator could be exacerbated by tamsulosin and result in putting the subject at risk of injury.
* Prior medical history or evidence of prostate cancer (e.g., positive biopsy, or suspicious ultrasound, or suspicious digital rectal examination (DRE)). Subjects with suspicious ultrasound or DRE who have had a negative biopsy within the preceding 6 months and stable prostate specific antigen (PSA) are eligible for the study. The investigator should make every appropriate effort to exclude the possibility of prostate cancer, including consideration of prostate biopsy in any subject with a known abnormal PSA.
* History of Breast cancer or clinical breast examination finding suggestive of malignancy Malignancy within the past five years, except for basal cell carcinoma of the skin.

Subjects with a prior malignancy who have had no evidence of disease for at least the past 5 years are eligible.

* History of any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions that could interfere with a subject's safety, or interfere with the subject's ability to follow indications or study procedures, or the interpretation of study results or obtaining informed consent or compliance to study procedures in the opinion of the Investigator or GSK Medical Monitor.
* History of myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident prior to Screening visit; or diabetes or peptic ulcer disease which is uncontrolled by medical management.
* Unable to refrain from the use of strong CYP3A4 inhibitors (e.g. ketoconazole) and/or strong CYP2D6 inhibitors (e.g. paroxetine) throughout the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-10-25 (Actual); Primary Completion 2014-01-22 (Actual); Study Completion 2014-01-22 (Actual)

PRIMARY OUTCOMES:
To evaluate the pharmacokinetics of dutasteride and tamsulosin when dosed alone and in combination | Pre-dose (within 10 minutes of the dutasteride administration), 0.25, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 48 and 72 hours post dose.Pre-dose (within 10 minutes of tamsulosin administration) on Day 1, Day 2 and Day 3 and pre-dose, 0.25, 0.5, 1, 2, 3, 4, 6,
  Serum dutasteride AUC (0-t), Cmax, tmax, following 0.5mg single dose administration with and without tamsulosin 0.2mg q24h. Serum tamsulosin AUC(0-τ), Cmax, tmax, Cτ and CL/F following 0.2mg q24h administration with and without dutasteride 0.5mg single dose.

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of dutasteride and tamsulosin when administered alone and in combination. | 11 Weeks
  AEs, SAEs, concurrent medication, changes in clinical laboratory values, ECG, and vital signs assessments.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 200254 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/200254?search=study&study_ids=200254#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200254 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register